CLINICAL TRIAL: NCT05478772
Title: A Phase 1, Open-Label, Fixed-Sequence, Drug-Drug Interaction Study to Evaluate the Effect of Multiple Doses of Fluconazole, a CYP3A4 and CYP2C9 Inhibitor, on the Pharmacokinetics of CTP-543 in Healthy Subjects
Brief Title: Study to Evaluate Multiple Doses of Fluconazole, a CYP3A4 and CYP2C9 Inhibitor, on the Pharmacokinetics of CTP-543 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP543.1015
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Health Volunteers
Keywords: CTP-543
MeSH Terms: interventions — Fluconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTP-543 and Fluconazole Treatment (Experimental): On Day 1, each subject will receive a single oral dose of 12 mg CTP-543. Following a washout on Day 2, each subject will receive an oral dose of 200 mg fluconazole once daily on Days 3 through to Day 8. On Day 7, approximately 1 hour after the 200 mg dose of fluconazole, each subject will receive a single oral dose of 12 mg CTP-543.
  Interventions: Drug: CTP-543; Drug: Fluconazole

INTERVENTIONS:
Drug: CTP-543 — 12 mg on Day 1 and Day 7
Drug: Fluconazole — 200 mg once daily on Days 3 through to Day 8

SUMMARY:
A single center, Phase 1, open-label, fixed-sequence, drug-drug interaction study to evaluate the effect of multiple doses of Fluconazole, a CYP3A4 and CYP2C9 inhibitor, on the pharmacokinetics (PK) of CTP-543 in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, aged 18-60 inclusive
* Non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at screening
* If of reproductive age, willing and able to use a medically highly effective form of birth control 4 weeks prior to first dose, during the study and for 30 days following last dose of study medication.
* Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease
* History or presence of alcohol or drug abuse within the past 2 years
* History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds
* Presence or history of significant gastrointestinal, liver or kidney disease, or any other condition that is known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
* History of prolonged QT syndrome or a QTc interval with Fridericia's correction (QTcF) > 450 msec for males or QTcF > 470 msec for females at Screening visit or prior to the first dosing
* Abnormal liver function at Screening
* Females who are nursing, pregnant, or planning to become pregnant while in the study, and for 30 days after last dose of study drug
* Positive results for coronavirus infection (COVID-19) at Screening or check-in
* Positive drug or alcohol results at Screening or check-in
* Positive results at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* Vaccination with a live attenuated vaccine up to 6 weeks prior to dosing. Live vaccines include (but are not limited to) the measles, mumps, and rubella (MMR) vaccine; intranasal flu vaccine; and Zostavax for herpes zoster

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-08-06 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
  Maximum observed concentration
Tmax | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
  Time to reach maximum observed concentration
λz | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
  Terminal elimination rate constant
t1/2 | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
  Apparent terminal half-life
AUC0-tlast | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
  Area under the concentration-time curve from time 0 to the time of the last observed/measured non-zero concentration
AUC0-inf | Pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36 and 48 hours post-dose
  Area under the concentration-time curve from time 0 extrapolated to infinity

SECONDARY OUTCOMES:
Assessment of Safety and Tolerability following administration of CTP-543 | Continuous from screening (within 21 days prior to Day 1) through Discharge (approximately 7 days after last study drug administration)
  Number of adverse events, including abnormal clinical laboratory findings, abnormal physical examinations, abnormal ECGs and abnormal vital signs tabulated for each subject

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, LLC, Miami, Florida, United States